CLINICAL TRIAL: NCT06849206
Title: Pennington Generation Cohort
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Professor, Pennington Biomedical Research Center
Other Study IDs: 2024-036
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity Prevention
Keywords: physical activity; obesity; diet; nutrition; families
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Pennington Generation Cohort is an observational study comprised of Louisiana families. Families will be assessed at baseline for a variety of traits and behaviors, and then followed up over time to try to understand the role of lifestyle and the environment on the risk of developing obesity and other health outcomes.

DETAILED DESCRIPTION:
Pennington Biomedical's Greaux Healthy initiative partners with communities to grow healthier generations by expanding the access and reach of Pennington Biomedical's evidence-based practices for the prevention and treatment of childhood obesity. As part of Greaux Healthy, the Pennington Generation Cohort will help evaluate the impact of the program. A sample of up to 1,500 children and adolescents and their families will be recruited from throughout Louisiana. An initial physical exam will establish a baseline for each family with respect to lifestyle behaviors, genetics, and body size/composition. This longitudinal cohort will also assess the association between participation in several childhood obesity prevention and treatment programs and subsequent obesity and related health outcomes. Members of the longitudinal cohort will be followed in the future through clinical visits, questionnaires, and through optional linkages to electronic medical records and administrative databases such as the National Death Index, Social Security Death Master File, and health registry data.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents, and young adults (birth through age 24 years) and their nuclear family members* and adults age 25+ who are expectant parents or are trying to conceive
* Self-reported resident of Louisiana
* Ability to understand instructions and complete all study procedures
* Able to provide informed consent (adults aged over 18 years)
* Able to provide assent (children 9 to 17 years)
* Able to communicate (oral and written) in English

Exclusion Criteria:

* Discretion of the Medical Monitor or Principal Investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults of child-bearing age who are planning to become pregnant, expectant parents, as well as children, adolescents, and young adults and their nuclear family members will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2045-02-24 (Estimated); Study Completion 2045-02-24 (Estimated)

PRIMARY OUTCOMES:
Obesity | From enrollment up to 20 years of follow-up.
  The development of obesity, defined using BMI z-scores during childhood, and BMI during adulthood.

SECONDARY OUTCOMES:
Weight change | From enrollment up to 20 years of follow-up.
  Change in body weight.
Mortality | From enrollment up to 20 years of follow-up..
  Data from the Pennington Generation Prospective Cohort will be prospectively linked to the National Death Index for the ascertainment of mortality.
Cancer incidence | From enrollment up to 20 years of follow-up..
  Data from the Pennington Generation Prospective Cohort will be prospectively linked to the Louisiana Tumor Registry for the ascertainment of incident cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified individual-level dataset will be made available to researchers making a reasonable request to the principal investigator.
Supporting Information: Study Protocol
Time Frame: Data will be made available 1 year after publication of the primary outcomes manuscript.
Access Criteria: Upon reasonable request to the principal investigator and in alignment with the goals of the IRB-approved protocol.